CLINICAL TRIAL: NCT07396727
Title: Health Professionals' Perceptions of the Subconscious Effects of Intraoperative Conversations in Patients: A Questionnaire-Based Study
Brief Title: Subconscious Effects of Intraoperative Speech: Health Professionals' Perceptions
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine OZCAN, Principal Investigator, Başakşehir Çam & Sakura City Hospital
Other Study IDs: AWAKE2025
Record Dates: First submitted 2025-09-26; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intraoperative Awareness; Anesthesia, General; Consciousness
Keywords: Anesthesia, General; Intraoperative Awareness; Consciousness; Health Personnel; Operating Rooms
MeSH Terms: conditions — Intraoperative Awareness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operating Room Health Professionals: Anesthesiologists, anesthesia residents, anesthesia technicians, surgeons, surgical residents, and operating room nurses working actively in operating rooms across Turkey.
  Interventions: Other: Questionnaire / Survey

INTERVENTIONS:
Other: Questionnaire / Survey — An anonymous, structured 19-item online questionnaire (Google Forms) administered to operating room health professionals, including anesthesiologists, anesthesia residents, anesthesia technicians, surgeons, surgical residents, and operating room nurses. The survey collects demographic information, awareness, attitudes, and perceptions regarding the potential subconscious effects of intraoperative conversations.

SUMMARY:
This observational, questionnaire-based study aims to evaluate health professionals' perceptions regarding the potential subconscious effects of intraoperative conversations on patients. Although intraoperative awareness is rare, neuroscientific evidence suggests that unconscious perception of auditory stimuli under anesthesia may influence postoperative psychological outcomes. An anonymous 19-item online survey will be distributed to anesthesiologists, anesthesia residents, anesthesia technicians, surgeons, surgical residents, and operating room nurses across Turkey. Data will be collected via Google Forms, with voluntary participation and informed consent. Statistical analysis will include descriptive and comparative methods to assess differences across professional groups and experience levels.

DETAILED DESCRIPTION:
Intraoperative awareness refers to conscious or subconscious perception during general anesthesia. Although its clinical incidence is rare, previous studies using EEG, fMRI, and neurocognitive methods have shown that auditory stimuli presented during anesthesia can leave subconscious traces and may influence postoperative psychological well-being, trust in healthcare, and anxiety levels.This study aims to explore health professionals' knowledge, awareness, and attitudes regarding the potential subconscious effects of intraoperative conversations. The research is designed as a multicenter, observational, cross-sectional, questionnaire-based study. A 19-item anonymous online survey will be distributed through professional networks, social media, and institutional mailing lists. Target participants include anesthesiologists, anesthesia residents, anesthesia technicians, surgeons, surgical residents, and operating room nurses actively working in operating rooms across Turkey. The primary objective is to evaluate the awareness level of healthcare professionals on the potential subconscious effects of intraoperative speech. Secondary objectives include identifying differences between professional groups, years of experience, and demographic factors. No intervention or treatment is involved, and no patient participation is required. Participation is voluntary and anonymous, with informed consent obtained at the beginning of the online survey. The anticipated sample size is a minimum of 150 participants to allow meaningful subgroup comparisons. Data will be collected via Google Forms and analyzed using SPSS software. Descriptive statistics, group comparisons (t-test, ANOVA, Mann-Whitney U, Kruskal-Wallis), and chi-square tests will be performed. If sufficient sample size is achieved, correlation and regression analyses may also be conducted. This study is expected to provide valuable insights into the level of professional awareness and ethical considerations regarding intraoperative communication, potentially contributing to the development of training strategies to reduce intraoperative awareness risks and improve patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Currently working in an operating room environment in Turkey (e.g., anesthesiologist, anesthesia resident, anesthesia technician, surgeon, surgical resident, operating room nurse)
* Access to the internet and ability to complete an online questionnaire
* Willingness to participate voluntarily and provide informed consent via the online form

Exclusion Criteria:

* Individuals younger than 18 years
* Healthcare personnel not directly working in the operating room environment.
* Participants who provide incomplete, misleading, or random responses in the questionnaire
* Individuals who do not provide informed consent at the beginning of the online survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Operating room health professionals in Turkey, including anesthesiologists, anesthesia residents, anesthesia technicians, surgeons, surgical residents, and operating room nurses. Participation is voluntary and limited to individuals aged 18 years and older who provide informed consent to complete the online questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Awareness and Perceptions of Health Professionals Regarding Subconscious Effects of Intraoperative Conversations | At survey completion (single time point) during the 1-month data collection period
  Evaluated through responses to a 19-item anonymous online questionnaire. Measured parameters include knowledge of intraoperative awareness, beliefs about subconscious auditory perception under anesthesia, and attitudes toward ethical and professional considerations. Responses are assessed using Likert scales, categorical questions, and descriptive statistics.

SECONDARY OUTCOMES:
Differences in Awareness Across Professional Groups | At survey completion (single time point) during the 1-month data collection period
  The evaluation was based on responses to a 19-item anonymous online survey. Comparison of perceptions regarding patient awareness during anesthesia among anesthesiologists, anesthesia assistants, anesthesia technicians, surgeons, surgical assistants, and operating room nurses.
Correlation between Age and Awareness/Professional Attitude Score | At survey completion (single time point) during the 1-month data collection period
  Association between participant age (years) and the composite awareness/professional attitude score measured by the online questionnaire.
Support for Training and Ethical Guidelines | At survey completion (single time point) during the 1-month data collection period
  Evaluated through responses to a 19-item anonymous online questionnaire. Proportion of participants endorsing the need for training programs and ethical standards addressing intraoperative communication.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Ozcan, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Başakşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study collects anonymous survey responses only. No individual participant data (IPD) will be shared.

REFERENCES:
- [Background] Fu VX, Sleurink KJ, Janssen JC, Wijnhoven BPL, Jeekel J, Klimek M. Perception of auditory stimuli during general anesthesia and its effects on patient outcomes: a systematic review and meta-analysis. Can J Anaesth. 2021 Aug;68(8):1231-1253. doi: 10.1007/s12630-021-02015-0. Epub 2021 May 19. PMID 34013463
- [Background] Kim KM, Bang JY, Choi BM, Noh GJ. Assessment of explicit and implicit memories during remimazolam anaesthesia using the process dissociation procedure: A prospective cohort study. Eur J Anaesthesiol. 2023 Nov 1;40(11):833-840. doi: 10.1097/EJA.0000000000001904. Epub 2023 Sep 25. PMID 37747426
- [Background] Han L, Purger DA, Eagleman SL, Halpern CH, Buch V, Gaston SM, Razavi B, Meador K, Drover DR. Deep learning models using intracranial and scalp EEG for predicting sedation level during emergence from anaesthesia. BJA Open. 2024 Oct 12;12:100347. doi: 10.1016/j.bjao.2024.100347. eCollection 2024 Dec. PMID 40018289
- [Background] Jang H, Mashour GA, Hudetz AG, Huang Z. Measuring the dynamic balance of integration and segregation underlying consciousness, anesthesia, and sleep. bioRxiv [Preprint]. 2024 Apr 15:2024.04.12.589265. doi: 10.1101/2024.04.12.589265. PMID 38659759